CLINICAL TRIAL: NCT05920798
Title: MC220601, Folate Receptor Alpha Dendritic Cells (FRαDCs) Plus Pembrolizumab for Patients With Advanced Stage Ovarian Cancer (FRAPPE)
Brief Title: Vaccine Therapy Plus Pembrolizumab in Treating Advanced Ovarian, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Acronym: FRAPPE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: NanoPass Technologies Ltd (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC220601; NCI-2023-03999 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-000139 (Other: Mayo Clinic Institutional Review Board); MC220601 (Other: Mayo Clinic); R01CA276313 (NIH)
Record Dates: First submitted 2023-06-09; First posted 2023-06-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fallopian Tube Carcinosarcoma; Primary Peritoneal Carcinosarcoma; Recurrent Fallopian Tube Carcinoma; Recurrent Fallopian Tube Clear Cell Adenocarcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Fallopian Tube High Grade Serous Adenocarcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Carcinosarcoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Clear Cell Adenocarcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Carcinosarcoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (apheresis, FRalphaDC, pembrolizumab) (Experimental): Patients undergo apheresis for multi-epitope folate receptor alpha-loaded dendritic cell vaccine manufacturing on study. Patients then receive multi-epitope folate receptor alpha-loaded dendritic cell vaccine ID on day 1 of cycles 1-5 and pembrolizumab IV over 30 minutes on day 1 of cycles 1-8. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patient then receive multi-epitope folate receptor alpha-loaded dendritic cell vaccine ID on day 1 of odd cycles and pembrolizumab IV over 30 minutes on day 1 of remaining cycles. Cycles repeat every 42 days for up to cycle 22 in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI as well as blood sample collection throughout the trial. Patients undergo biopsy on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine; Biological: Pembrolizumab; Procedure: Pheresis

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Multi-epitope Folate Receptor Alpha-loaded Dendritic Cell Vaccine — Given ID
  Other Names: FRaDC Vaccine; FRalphaDC Vaccine
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis

SUMMARY:
This phase I/II trial tests the safety, side effects, best dose, and effectiveness of multi-epitope folate receptor alpha-loaded dendritic cell vaccine (FRalphaDC) with pembrolizumab in treating patients with ovarian, fallopian tube, or primary peritoneal cancer (collectively known as ovarian cancer) that that has come back (after a period of improvement) (recurrent). Ovarian cancer is the most lethal gynecologic malignancy in the United States. While the majority of patients achieve a remission from ovarian cancer with the combination of aggressive cytoreductive surgery and cytotoxic chemotherapy, over 80% of patients develop recurrence within 3 years of completion of treatment. Additional treatments are needed for recurrence, but the standard treatment modalities are non-curative in nature due to the development of drug resistance. As such, there is a great unmet need for treatment strategies that utilize new mechanisms to which drug resistance does not develop. FRalphaDC is a dendritic cell vaccine that is made from the white blood cells collected from a procedure call apheresis. The white blood cells are treated to make dendritic cells, which will then be incubated with peptides, which are pieces of a protein known as "folate receptor alpha" (FRalpha), a protein that is found in high levels on ovarian cancer cells. Dendritic cell vaccines work by boosting the immune system (a system in the body that protect against infection) to recognize and destroy the tumor cells by targeting the FRalpha protein. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving FRalphaDC vaccine with pembrolizumab may be a safe and effective treatment for recurrent ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the combination of FRalphaDCs and pembrolizumab has an acceptable toxicity profile in patients with recurrent ovarian cancer (OC). (Phase I) II. To measure the confirmed objective response rate (ORR) to the combination of FRalphaDCs and pembrolizumab in patients with recurrent OC. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the disease control rate (DCR-percentage of patients achieving a complete response, partial response, or stable disease) of the combination of FRalphaDCs and pembrolizumab in patients with recurrent OC.

II. To estimate the duration of response (DoR) in patients with recurrent OC treated with the combination of FRalphaDCs and pembrolizumab.

III. To estimate the progression-free survival (PFS) of patients with recurrent OC treated with the combination of FRalphaDCs and pembrolizumab.

IV. To estimate the overall survival (OS) of patients with recurrent OC treated with the combination of FRalphaDCs and pembrolizumab.

2.25 To characterize the adverse event (AE) profile in patients with recurrent OC treated with the combination of FRalphaDCs and pembrolizumab.

CORRELATIVE OBJECTIVES:

I. To determine whether the combination of FRalphaDCs and pembrolizumab induces an increase in the frequency of FRalpha-specific IL-17-secreting T cells (Th17s) in patients with recurrent OC.

II. Characterize the T cell and antibody responses to FRalpha and assess the association between the emergence of immunity and recurrence-free (RFS).

III. To determine whether the combination of FRalphaDCs and pembrolizumab induces an increase in the frequency of FRalpha-specific IFNgamma-secreting T cells (Th1s) in patients with recurrent OC.

IV. To determine whether the combination of FRalphaDCs and pembrolizumab induces an increase in the frequency of FRalpha-specific IgG antibodies in patients with recurrent OC.

V. To determine whether the combination of FRalphaDCs and pembrolizumab induces changes in the immune microenvironment of ovarian tumors.

OUTLINE:

Patients undergo apheresis for multi-epitope folate receptor alpha-loaded dendritic cell vaccine manufacturing on study. Patients then receive multi-epitope folate receptor alpha-loaded dendritic cell vaccine intradermally (ID) on day 1 of cycles 1-5 and pembrolizumab intravenously (IV) over 30 minutes on day 1 of cycles 1-8. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patient then receive multi-epitope folate receptor alpha-loaded dendritic cell vaccine ID on day 1 of odd cycles and pembrolizumab IV over 30 minutes on day 1 of remaining cycles. Cycles repeat every 42 days for up to cycle 22 in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) as well as blood sample collection throughout the trial. Patients undergo biopsy on study.

Patients are followed up at 90 days after last dose, every 3 months until 24 months after registration or until progression of disease, and then every 6 months up to 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically confirmed recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer NOTE: Histologic confirmation of the primary tumor or recurrent tumor per pathology report is required. Eligible histotypes include high grade serous; endometrioid; and clear cell carcinoma, as these histotypes have high expression of FRalpha. Mixed carcinomas, including carcinosarcomas, with >= 50% of the tumor comprised of high grade serous; and/or endometrioid; and/or clear cell carcinoma are eligible
* Ovarian cancer (OC) recurrence - Platinum sensitivity/resistance

  * Platinum-refractory (defined as recurrence or progression of OC =< 30 days of the last dose of platinum-based chemotherapy)
  * Platinum-resistant (defined as recurrence or progression of OC between 31-180 days of the last dose of platinum-based chemotherapy)
  * Platinum-sensitive (defined as recurrence or progression >=181 days after the last dose of platinum-based chemotherapy).

NOTE: Any number of prior therapies or maintenance regimens for OC are allowed

* At least one of the following:

  * Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria AND/OR
  * CA-125-evaluable disease, as defined by the Gynecologic Cancer InterGroup (GCIG)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 8.5 g/dL (obtained =< 15 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 15 days prior to registration)
* Lymphocytes >= 0.3 x 10^9/L (obtained =< 15 days prior to registration)
* Monocytes >= 0.25 x 10^9/L (obtained =< 15 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless patient has a documented history of Gilbert's disease, then direct bilirubin must be =< ULN (obtained =< 15 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (obtained =< 15 days prior to registration)
* Creatinine clearance >= 30 mL/min per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation (obtained =< 15 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to provide mandatory blood and tissue specimens for correlative research
* Willing to provide archival tissue specimen for correlative research
* Willing to return to Mayo Clinic for follow-up (during the active monitoring phase of the study)
* Willing to undergo a tetanus vaccination (if not performed =< 365 days prior to registration)
* Willing to have a temporary central access line placed for apheresis, if needed

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic and teratogenic effects of which on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Prior treatment for ovarian cancer with an anti-PD-1 or anti-PD-L1 monoclonal antibody
* Treatment with IV anti-cancer therapy =< 3 weeks prior to registration or with oral anti-cancer therapy =< 1 week prior to registration NOTE: Since treatment will begin no sooner than 4 weeks after registration due to the need for apheresis and manufacturing of the FRαDC product, a "wash-out" period prior to registration will cause a gap of at least 5 weeks between the last anti-cancer treatment and initiation of protocol therapy
* Grade 2 or higher symptoms attributed to OC OR disease measuring > 5 cm in long axis (non-nodal lesions), or > 5 cm in short axis (nodal lesions) OR disease that, in the judgement of the treating investigator, is likely to become symptomatic in the next 8 weeks (ex. moderate ascites)

  * NOTE: Since patients will not receive therapy for cancer until 3-4 weeks after apheresis--which is potentially 6-8 weeks after registration --patients with symptomatic OC or an elevated tumor burden may experience significant progression prior starting therapy and should not be treated on this protocol).
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled human immunodeficiency virus (HIV) infection and/or HIV-infected patients with a history of Kaposi's sarcoma and/or multicentric Castleman disease.

  * NOTE: HIV-infected participants must have well-controlled HIV on anti-retroviral therapy (ART), defined as:

    * Participants on ART must have a CD4+ T-cell count ≥ 350 cells/mm^3 at the time of screening
    * Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV ribonucleic acid (RNA) level below 50 or the lower limit of quantification derivation technique (LLOQ) (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
    * It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months
    * Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (day 1) and agree to continue ART throughout the study
  * NOTE: No HIV testing is required unless mandated by local health authority
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active serious infections (e.g., pneumonia, sepsis) requiring systemic therapy
  * Current diagnosis or previous history of immune-related (non-infectious) pneumonitis or interstitial lung disease that requires or required steroids
  * Active autoimmune disease that required systemic treatment other than replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroids) =< 2 years prior to registration
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Concurrent active hepatitis B [defined as hepatitis B surface antigen (HBsAg) positive and/or detectable hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ] and Hepatitis C virus [defined as anti-hepatitis C virus (HCV) antibody (Ab) positive and detectable HCV RNA] infection. EXCEPTIONS:

    * For patients with evidence of hepatitis B virus (HBV) infection (HBsAg positive), patients must have completed at least 4 weeks of hepatitis B virus (HBV) antiviral therapy and the HBV viral load must be undetectable at the time of registration

      * NOTE: Patients should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention
    * Patients with a history of hepatitis C virus (HCV) are eligible if they have an undetectable HCV viral load.

      * NOTE: Patients must have completed curative anti-viral treatment >= 4 weeks prior to registration
  * NOTE: Patients without symptoms or prior history do not require testing prior to registration unless mandated by local health authority
* Other active malignancy either requiring palliative systemic therapy =< 3 years prior to registration, or likely to require treatment in the next 2 years EXCEPTIONS: Patients with non-melanotic skin cancer, papillary thyroid cancer not requiring therapy or carcinoma-in-situ are eligible for this trial. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias NOTE: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Treatment with systemic immunosuppressive medication (including, but not limited to, prednisone >10 mg/day or equivalent, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF]-alpha agents) =< 7 days prior to registration, or anticipation of need for systemic immunosuppressive medication during the course of the study NOTE: Patients who have received acute, low-dose systemic steroids (=< 10 mg/day oral prednisone or equivalent) prior to registration or a one-time pulse dose of systemic immunosuppressant medication (e.g., =< 48 hours of corticosteroids for a contrast allergy) are eligible for the study NOTE: The use of inhaled corticosteroids for chronic obstructive pulmonary disease or asthma, mineralocorticoids (e.g., fludrocortisone), or low-dose corticosteroids for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of allogeneic stem cell transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Determine whether the combination of FRαDCs and pembrolizumab has an acceptable toxicity profile. | Up to 21 days
  Three patients will be enrolled to starting dose (dose level 1) and enrollment will pause until each of the first 3 patients have completed cycle 1 of therapy. If zero or one of first 3 patients develops a dose limiting toxicity (DLT) during cycle 1, 3 more patients will be enrolled to dose level 1. If observe at most 1 DLT in the first 6 patients at dose level 1, it will be considered safe and will continue in phase II of trial. If 2 or more of the first 6 patients develop a DLT during cycle 1 for dose level 1, then enrollment will stop and dose level will be decreased. Additional patients will be enrolled in cohorts of 3 to that decreased dose level. If zero or one DLT in the first 6 patients at dose level -1, it will be considered safe and will continue in phase II of trial. Otherwise, if observe 2 or more DLTs in the first 6 patients of dose level -1, enrollment will stop until the Study Team adjusts the treatment plan with input from the Data Safety Monitoring Board.
Confirm objective response rate (ORR) | Up to 5 years
  Defined as the proportion of patients with a complete response (CR) or partial response (PR). If at least 7 confirmed responses are observed in the first 32 eligible patients (22%), the combination treatment will be considered worthy of further investigation.

SECONDARY OUTCOMES:
Disease control rate | Up to 5 years
  Defined as the proportion of patients with a complete response (CR),partial response (PR), or stable disease.
Duration of response | Up to 5 years
  Duration of response (DoR) is defined as the time from the first disease assessment showing a complete response (CR) or partial response (PR) until the date of either disease progression or death of any cause.
Progression free survival (PFS) | Up to 5 years
  PFS will be estimated using the Kaplan-Meier method. The date of progression will be the date on which progressive disease is first detected, even if the patient does not immediately come off study.
Overall survival (OS) | Up to 5 years
  OS will be estimated using the Kaplan-Meier method. OS is defined as the time from study entry to death from any cause.
Incidence of adverse events | Up to 5 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials